CLINICAL TRIAL: NCT03514589
Title: NeSST2: A Multi-stage Clinical Study to Develop a Non-invasive Short Synacthen Test (SST)
Brief Title: NeSST2: The Development of a Noninvasive Short Synacthen Test
Acronym: NeSST2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH/12/043
Record Dates: First submitted 2015-12-21; First posted 2018-05-02 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Adrenal Suppression
MeSH Terms: interventions — Cosyntropin; adrenocorticotropin zinc

STUDY DESIGN:
Intervention Model Description: Current stage is stage 3 (Sept 2023), an open label study of nasal Synacthen in healthy children aged 0-18 to derived normative reference data.
  Previous stages:
  1a: 12 healthy adult males, 4 arms (dose selection studying nasal synacthen 100 mcg + chitosan, 500 mcg and 500 mcg + chitosan against 1mcg IV Synacthen)
  1b: 6 healthy adult males 1 arm (repeatability: two further 500 mcg + chitosan visits)
  1c: 12 healthy adult males 3 arms (dose rangign study: 500 mcg + chitosan, 1mg + chitosan against 250 mcg IV Synacthen comparator) 2: Healthy children aged 2-15 (500 mcg + chitosan, against 145 mcg/m2 IV Synacthen comparator)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): 250 mcg IV synacthen
  Interventions: Drug: nasal Tetracosactide
- Arm 2 (Experimental): Nasal Synacthen
  Interventions: Drug: IV tetracosactide

INTERVENTIONS:
Drug: nasal Tetracosactide — Bioavailability of nasal synacthen compared to IV comparator
  Other Names: cosyntropin; Synacthen
  Arms: Arm 1
Drug: IV tetracosactide — Bioavailability of nasal synacthen compared to IV comparator
  Other Names: cosyntropin; synacthen
  Arms: Arm 2

SUMMARY:
Recently there has been concern about the effect of inhaled steroids, routinely used in the treatment of asthma, on the body's ability to produce its natural stress hormone cortisol. Failure of adequate cortisol production in times of stress e.g. illness, can result in serious illness or death. Patients receiving longterm steroid treatment may have reduced levels of cortisol and not be able to produce adequate amounts in times of need, a process called adrenal suppression. Initially it was thought that the absorption of inhaled steroids into the bloodstream would be too low to cause adrenal suppression however high profile deaths followed by a national survey revealed a number of fatal or near fatal cases of adrenal suppression. The vast majority of these were in children. Since then doctors have been encouraged to ensure that children on high doses of inhaled steroids carry a steroid alert card and that the ability of their adrenal glands to produce adequate amounts of cortisol is checked. However it is unknown what dose of inhaled steroids puts one at risk, whether age or gender affects one's risk and when to check the function of the adrenal gland.

The Short Synacthen Test (SST) investigates the ability of the body's adrenal glands to produce cortisol. Presently the SST requires intravenous (i.v) cannulation through which Synacthen is injected to stimulate the adrenal glands and multiple blood samples are collected to assess the response in terms of cortisol production. It is invasive, time consuming and unpleasant for the child. Our project aims to produce a noninvasive alternative to the current SST, with Synacthen given nasally and using saliva to measure the subsequent production of cortisol. A noninvasive test will allow us to establish the first normal ranges for children and determine which children with asthma are at risk of adrenal suppression.

DETAILED DESCRIPTION:
The success of the nasal administration of a novel formulation of Synacthen to adults was the first step in a work-stream, which aims to develop the clinical applicability of the non-invasive SST in addition to using it as an important research tool. The invasive nature of the current diagnostic test makes large cohort research impracticable. Having gained proof of concept with the initial study we will now go on to gained detailed pharmacokinetic information in adults with the IV comparator of the 250 mcg test in addition to the data already gained for the 1 mcg test. We will test two doses of nasal Synacthen. We will do intra-individual variation work also.

The next stage will then to be to perform pharmacokinetic validation of the nasal Synacthen plus chitosan dose in twenty children in order to establish that the chosen dose, peak cortisol response, bioavailability and pharmacokinetics are similar in the paediatric population. This will require 40 visits to our Childrens' Clinical Research Facility.

In order to obtain the quality of pharmacokinetic data required for commercial regulatory approvals an improved Synacthen assay is required. This work is ongoing in collaboration with ACTH assay experts at the University of Manchester.

ELIGIBILITY:
Inclusion Criteria:

Stage 1b+c:

• Healthy, male volunteers aged between 18-64 with none of the exclusion criteria listed below.

Stage 2:

• Healthy children of either sex, aged between 2 and 15 years (up to their 16th birthday) with none of the exclusion criteria listed below.

Stage 3:

• Healthy children of both sexes, aged between 0-18 years without exclusion criteria 1,2,3,5,6,7,8,9,10,11,12,14 listed below.

Stage 4:

• Asthmatic children of both sexes, aged between 6 months and 15 years, prescribed regular inhaled corticosteroids and without exclusion criteria 1,5,9,10,11,12, and 14 listed below.

Exclusion Criteria:

1. Past or present history of an endocrinopathy (all stages)
2. Past or present history of asthma (stages 1b+c,2,3)
3. Past or present history of allergic rhinitis (stages 1b+c,2,3)
4. Past or present history of peptic ulcer disease/GI bleed/significant dyspepsia (stages 1b+c,2)
5. Past history of intra-cranial or renal/adrenal pathology (all stages)
6. Presently on any medication (stages 1b+c,2,3)
7. Presently, or within the last 3 months, been prescribed any type of corticosteroid (oral, inhaled, nasal, rectal, intravenous, intramuscular, intra-articular, intra-ocular, topical) (stages 1b+c,2,3)
8. Ever been prescribed a prolonged course of oral corticosteroids (more than 1 month) (stages 1b+c,2,3)
9. Previous adverse reaction (including mild hypersensitivity) to ACTH or Synacthen (all stages)
10. Previous severe allergic reaction or anaphylaxis (all stages)
11. Coryzal symptoms within the last week (and will be asked to report any new symptoms occurring within 24 hours of the test) (all stages)
12. Current smoker (all stages)
13. Body Mass Index less than 18.5 or more than 30kg/m2 (stages 1b+c) outside 3rd to 97th centiles for ages and sex (stage 2)
14. Currently pregnant (stages 2,3,4)
15. Currently anaemic (stages 1b+c,2)

Ages: 6 Months to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-10-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Peak plasma cortisol concentration (Cmax) | 6 months
  Peak plasma cortisol following synacthen
Time of peak plasma cortisol concentration (Tmax) | 6 months
  Time of Cmax
Bioavailability of nasal Synacthen (compared to IV Synacthen) | 6 months
  Proportion of synacthen measurable in blood following administration (IV or nasal) and so is able to have an active effect.
Area under the curve for plasma Synacthen (nasal compared to IV) | 6 months
  Total exposure to synacthen
Area under the curve for plasma cortisol (nasal compared to IV) | 6 months
  Total exposure to plasma cortisol following synacthen

SECONDARY OUTCOMES:
Tolerability and acceptability of nasal Synacthen test | Course of the study (2.5 years)
  Questionnaire answers to questions on tolerability and acceptability of nasal Synacthen test. Safety data
Correlation of plasma cortisol with salivary cortisol | 6 months
  relationship of peak plasma cortisol and peak salivary cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Elder, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom

IPD SHARING:
Plan to Share IPD: No